CLINICAL TRIAL: NCT06666374
Title: Evaluating the Effectiveness and Persistence of an Oral Health Literacy Intervention on Oral Health Behaviors and Plaque Reduction in Orthodontic Patients: a Randomized Controlled Trial
Brief Title: Effectiveness of an Oral Health Literacy Intervention on Oral Health Behaviors and Plaque Index in Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Srinakharinwirot University (Other)
Responsible Party: Principal Investigator, Neeranart Thirasupa, Program director of Residency training program in Orthodontics, Srinakharinwirot University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 005/2566
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Dental Plaque; Periodontal Diseases; Oral Health Behavior Change
Keywords: Oral health literacy; Self-efficacy; Experiential learning; Oral health intervention; Oral health behavior; Plaque index
MeSH Terms: conditions — Dental Plaque; Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OHL Program (Experimental): This program used OHL as its core structure and incorporated elements of experiential learning and self-efficacy to enhance patient engagement and understanding.
  Interventions: Behavioral: OHL program
- Traditional program (Active Comparator): Patients acquired traditional oral health instruction from another dental professional, which primarily focused on providing information without the OHL components, self-efficacy strategies, or the interactive elements of the intervention program.
  Interventions: Behavioral: Traditional program

INTERVENTIONS:
Behavioral: OHL program — This program used OHL as its core structure and incorporated elements of experiential learning and self-efficacy to enhance patient engagement and understanding. The program comprised seven steps designed to guide patients through key aspects of oral health care, enabling them to progressively build their skills and confidence. These steps included personalized education on oral health, hands-on practice of proper oral hygiene techniques, self-assessment exercises, and strategies for overcoming barriers to good oral health.
  Other Names: OHL-OHI
  Arms: OHL Program
Behavioral: Traditional program — Program primarily focused on providing information without the OHL components, self-efficacy strategies, or the interactive elements of the intervention program.
  Other Names: Trad-OHI
  Arms: Traditional program

SUMMARY:
This study aims to evaluate the effectiveness of a novel psychologic-based oral health instruction program (OHL program) by comparing oral health behaviors (OHB) and plaque index (PI) scores between intervention and control groups at three key time points-pre-intervention, post-intervention, and follow-up-enabling a comprehensive assessment of the intervention's impact and and persistence over time. The study hypothesizes that (1) the OHL program will lead to greater improvements in OHL compared to a traditional control group and (2) these effects will be sustained through the follow-up period.

Participants in the intervention group received the OHL program, while those in the control group received traditional oral hygiene instruction. Both groups had data collected at baseline, post-intervention, and at a 3-week follow-up.

DETAILED DESCRIPTION:
The outcomes were oral health behavior (OHB) and plaque index (PI), compared at three time points: baseline (initial), post-intervention (final), and at a 3-week follow-up. Additionally, as a manipulation check, oral health literacy (OHL) levels were assessed at all three intervals.

Demographic information, OHL, and OHB were measured using standardized questionnaires from previous research. The 31-item OHL scale assessed five elements: 1) access, 2) understanding, 3) evaluation, 4) application, and 5) communication of oral health information and services. A 14-item scale evaluated OHB across three domains: 1) oral hygiene practices, 2) dietary choices, and 3) utilization of dental services.

In addition, clinical assessments of plaque were conducted using the Silness and Löe plaque index (PI, 1964). Plaque was evaluated on four surfaces of each tooth (mesial, distal, buccal, and lingual) using a WHO probe. Scores ranged from 0 to 3, reflecting the absence to a large amount of plaque accumulation, based on their established criteria. A single oral examiner recorded the plaque scores for each surface, and the average score for each tooth was calculated. The total score was then summed and divided by the total number of teeth examined, providing an overall plaque index for each individual. There were no outcome changes after trial commencement.

ELIGIBILITY:
Inclusion Criteria:

* participants undergoing fixed orthodontic treatment, free from non-communicable chronic diseases (such as diabetes mellitus, hypertension, and heart disease), capable of reading, writing, and providing informed consent, and willing to participate in the oral health program.

Exclusion Criteria:

* reluctance to provide health information, inability to complete assessments, or withdrawal from the program at any stage.

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Oral health behavior | Outcomes were measured at baseline, post-intervention, and at a 3-week follow-up, with a total study duration averaging 3 months.
  Oral hygiene care, Dietary choice, Dental visit
PI | Outcomes were measured at baseline, post-intervention, and at a 3-week follow-up, with a total study duration averaging 3 months.
  Plaque index score

SECONDARY OUTCOMES:
OHL | Outcomes were measured at baseline, post-intervention, and at a 3-week follow-up, with a total study duration averaging 3 months.
  Oral health literacy

CONTACTS AND LOCATIONS:
Locations (1):
- HRH Princess Maha Chakri Sirindhorn Medical Center, Nakhon Nayok, Changwat Nakhon Nayok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 1.5 years after the publication of results
Access Criteria: Permitted researchers will be able to access the IPD and supporting information. They will be allowed to receive the Study Protocol and Statistical Analysis Plan (SAP). Researchers must request permission from me first.